CLINICAL TRIAL: NCT01281137
Title: SOLE Estrogen Substudy (SOLE-EST) - Investigating Changes in Estrogen Levels and Grip Strength for Patients Participating in the SOLE Trial
Brief Title: Study of Changes in Estrogen Levels and Grip Strength in Postmenopausal Women Who Have Received 4 to 6 Years of Hormone Therapy for Breast Cancer and Are Currently Receiving Letrozole on Clinical Trial IBCSG-35-07
Acronym: SOLE-EST
Status: Completed | Type: Observational
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: CDR0000692740; IBCSG-35-07-SUBSTUDY (Other: IBCSG); BIG-1-07-SUBSTUDY (Other: Breast International Group); 2007-001370-88 (EudraCT Number); EU-21101
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood,
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: polymorphism analysis — SNPs will be genotyped in whole blood samples taken at baseline.
Other: laboratory biomarker analysis — Biomarkers will be assessed in blood and serum samples at different time points.
Procedure: quality-of-life assessment — Quality of life will be assessed using the Breast Cancer Prevention Trial (BCPT) Symptom Scales and the IBCSG Trial 35-07 QL Form.

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving treatment for cancer may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying changes in estrogen levels and grip strength in postmenopausal women who have received 4 to 6 years of hormone therapy for breast cancer and are currently receiving letrozole on clinical trial IBCSG-35-07.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the serum level of estrogens (Estradiol [E2], Estrone [E1], and Estrone Sulphate [E1S] and sex hormone binding globulin [SHBG]) in postmenopausal women with prior endocrine-responsive, node-positive, resectable breast cancer completing 4 to 6 years of adjuvant endocrine therapy and enrolled on clinical trial IBCSG-35-07 receiving letrozole.
* To determine the degree of recovery of E2, E1, and E1S during the 3-month letrozole-off gap.

Secondary

* To determine the association between estrogen level changes and the clinical outcomes of toxicity and quality of life.
* To determine the effect of prior adjuvant endocrine therapy, age, body mass index, and type of menopause on estrogen levels.
* To determine the variability of estrogen level changes and its association with germline single nucleotide polymorphisms.
* To examine changes in grip-strength score.

OUTLINE: This is a multicenter study.

All patients undergo blood sample collection at baseline for the analysis of single nucleotide polymorphisms, after randomization on clinical trial IBCSG-35-07 and prior to the beginning treatment on IBCSG-35-07. Patients also undergo serum collection at baseline and at 9, 10.5, and 12 months for the analysis of estrogen levels and sex hormone binding globulins. Patients undergo measurement of grip strength at baseline and at 9 and 12 months. Samples may be banked for future research studies.

Patients complete quality-of-life questionnaires (Breast Cancer Prevention Trial [BCPT] Symptom Scales on Form 35-PRS and IBCSG Trial 35-07 QL Form) periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously diagnosed with breast cancer

  * Endocrine-responsive, node-positive, resectable disease
* Disease-free following 4-6 years of prior adjuvant endocrine therapy with selective estrogen-receptor modulators and/or aromatase inhibitors
* Patient must be currently enrolled on clinical trial IBCSG-35-07 as well as the Quality-of-Life substudy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Postmenopausal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients randomized to the SOLE trial (IBCSG 35-07) and participate in the Quality of Life substudy.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacquie Chirgwin, MD, Study Chair — Box Hill Hospital; Guy Jerusalem, MD, PhD, Study Chair — CHU Liege - Domaine Universitaire du Sart Tilman
Locations (2):
- Box Hill Hospital, Box Hill, Victoria, Australia
- CHU Liege - Domaine Universitaire du Sart Tilman, Liège, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The phase 3 randomized, open-label Study of Letrozole Extension (SOLE) enrolled 4884 postmenopausal women between December 2007 and October 2012. Among them, 104 patients were enrolled in the SOLE Estrogen Substudy (SOLE-EST). SOLE was a multinational study performed in 240 centers of the Breast International Group-affiliated cooperative groups in 22 countries.
Pre-assignment Details: There were 104 patients enrolled during the active period (25 continuous letrozole, 79 intermittent letrozole). Blood samples were obtained from 103 patients at baseline. For the longitudinal analysis, patients (N=90) were included if they had at least one post-baseline sample. At 9, 10.5, and 12 months, 85 (21 continuous, 64 intermittent), 84 (20 continuous, 64 intermittent) and 81 (19 continuous, 62 intermittent), patients, respectively, could be included in longitudinal analyses.
Groups:
- Continuous Letrozole Treatment Group; Intermittent Letrozole Treatment Group: The phase 3 randomized, open-label Study of Letrozole Extension (SOLE) enrolled 4884 postmenopausal women between December 2007 and October 2012. Among them, 104 patients were enrolled in the SOLE Estrogen Substudy (SOLE-EST).Patients were randomized 1:1 for SOLE and enrolled in 1:3 ratio for SOLE-EST between continuous letrozole (2.5 mg/day orally for 5 years) and intermittent letrozole treatment (2.5 mg/day during 9 months followed by a 3 month interruption in years 1-4 and then 2.5 mg/day during all year 5).
Period: Baseline Population
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Started | 25 | 79
Completed | 25 | 78
Not Completed | 0 | 1
Not completed — No samples assayed (excluded from all analyses) | 0 | 1
Period: Analysis Population (Baseline)
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Started (13 patients excluded from the longitudinal analyses, baseline sample only) | 25 | 78
Completed | 21 | 69
Not Completed | 4 | 9
Not completed — baseline sample only so excluded from longitudinal analysis | 4 | 9
Period: Analysis Population (9 Months)
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Started | 21 | 69
Completed | 21 | 64
Not Completed | 0 | 5
Not completed — 5 from the baseline analysis population did not have samples assayed for the analysis at month 9. | 0 | 5
Period: Analysis Population (10.5 Months)
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Started | 21 | 64
Completed | 20 | 64
Not Completed | 1 | 0
Not completed — 1 from the baseline analysis population did not have a sample assayed for analysis at month 10.5 | 1 | 0
Period: Analysis Population (12 Months)
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Started | 20 | 64
Completed | 19 | 62
Not Completed | 1 | 2
Not completed — 3 from the baseline analysis population did not have a sample assayed for analysis at month 12 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Postmenopausal woman with hormone receptor-positive, lymph node-positive, and operable breast cancer of any age were included in the study. They must have undergone local treatment and have completed 4-6 years of adjuvant endocrine therapy. At enrollment, they had to be clinically free of breast cancer without any evidence of recurrence. Patients were randomized 1:1 for SOLE and enrolled in 1:3 ratio for SOLE-EST.
Groups:
- Continuous Letrozole Treatment Group; Intermittent Letrozole Treatment Group: Patients were randomized 1:1 for SOLE and enrolled in 1:3 ratio for SOLE-EST between continuous letrozole (2.5 mg/day orally for 5 years) and intermittent letrozole treatment (2.5 mg/day during 9 months followed by a 3 month interruption in years 1-4 and then 2.5 mg/day during all year 5).
- Total: Total of all reporting groups
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group | Total
Number analyzed (Participants) | 25 | 78 | 103
Age, Customized [Count of Participants; unit: Participants]
  Age at randomization, years: <55 | 6 | 23 | 29
  Age at randomization, years: 55-59 | 6 | 13 | 19
  Age at randomization, years: 60-64 | 3 | 15 | 18
  Age at randomization, years: 65-69 | 5 | 12 | 17
  Age at randomization, years: ≥70 | 5 | 15 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 78 | 103
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) at randomization [Count of Participants; unit: Participants]
  Normal (<25) | 12 | 27 | 39
  Overweight (25-<30) | 7 | 31 | 38
  Obese (≥30) | 6 | 20 | 26
  Unknown | 0 | 0 | 0
Type of menopause [Count of Participants; unit: Participants]
  Bilateral oophorectomy | 4 | 22 | 26
  Chemotherapy-induced amenorrhea | 7 | 8 | 15
  Natural menopause before breast cancer diagnosis | 13 | 41 | 54
  Natural menopause since breast cancer diagnosis | 1 | 7 | 8
Last (most recent) type of prior endocrine therapy (ET) [Count of Participants; unit: Participants]
  Aromatase inhibitor (AI) | 23 | 72 | 95
  Selective estrogen receptor modulators (SERM) | 2 | 6 | 8
Duration of prior AI [Count of Participants; unit: Participants]
  <6 months | 2 | 5 | 7
  6 months - <2 years | 0 | 3 | 3
  2 - <3 years | 5 | 14 | 19
  3 - <4 years | 3 | 10 | 13
  ≥4 years | 15 | 46 | 61
  Unknown | 0 | 0 | 0
Duration from end of prior ET to randomization [Count of Participants; unit: Participants]
  ≤ 1 month | 20 | 61 | 81
  >1 month | 5 | 17 | 22

OUTCOME MEASURES:

1. Primary Outcome: Levels of Estrone (E1), Estradiol (E2), and Estrone Sulphate (E1S) Among Patients in the Longitudinal Analysis Population
Description: In SOLE-EST, levels of E1, E2, and E1S were summarized over time at 0 (baseline), 9, 10.5, and 12 months from randomization among patients in the longitudinal analysis population (N=90 with post-baseline sample).
Time Frame: 0 (baseline), 9, 10.5, and 12 months from randomization
Population: Longitudinal analysis group: There were 90/103 patients (21 continuous, 69 intermittent) who had baseline and one or more samples at 9, 10.5 and/or 12 months and could be included in analyses of hormone levels over time. At 9, 10.5, and 12 months, 85, 84, and 81, respectively, could be included in analyses of hormone levels over time.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Continuous Letrozole Treatment Group (Baseline, Month 0); Intermittent Letrozole Treatment Group (Baseline, Month 0); Continuous Letrozole Treatment Group (9 Months); Intermittent Letrozole Treatment Group (9 Months); Continuous Letrozole Treatment Group (10.5 Months); Intermittent Letrozole Treatment Group (10.5 Months); Continuous Letrozole Treatment Group (12 Months); Intermittent Letrozole Treatment Group (12 Months): There were 90/103 patients (21 continuous, 69 intermittent) who had baseline and one or more samples at 9, 10.5 and/or 12 months and could be included in analyses of hormone levels over time. At 9, 10.5, and 12 months, 85 (21 continuous, 64 intermittent), 84 (20 continuous, 64 intermittent), and 81 (19 continuous, 62 intermittent), patients, respectively, could be included in analyses of hormone levels over time.
Arm/Group | Continuous Letrozole Treatment Group (Baseline, Month 0) | Intermittent Letrozole Treatment Group (Baseline, Month 0) | Continuous Letrozole Treatment Group (9 Months) | Intermittent Letrozole Treatment Group (9 Months) | Continuous Letrozole Treatment Group (10.5 Months) | Intermittent Letrozole Treatment Group (10.5 Months) | Continuous Letrozole Treatment Group (12 Months) | Intermittent Letrozole Treatment Group (12 Months)
Number analyzed (Participants) | 21 | 69 | 21 | 64 | 20 | 64 | 19 | 62
pg/mL
  E1 | 12.4 [9.7 to 23.4] | 14.3 [5.8 to 26.1] | 4.8 [4.2 to 5.5] | 5.1 [4.3 to 5.8] | 4.7 [3.9 to 5.5] | 21.6 [15.4 to 29.7] | 5.1 [4.4 to 7.0] | 26.8 [18.5 to 35.7]
  E2 | 4.6 [3.3 to 7.3] | 4.7 [3.4 to 6.9] | 2.6 [2.2 to 4.0] | 3.2 [2.4 to 4.0] | 2.6 [2.0 to 3.7] | 6.7 [4.8 to 8.7] | 2.9 [2.3 to 4.0] | 7.3 [5.4 to 10.5]
  E1S: number analyzed (Participants) | 21 | 69 | 21 | 63 | 20 | 63 | 19 | 62
  E1S | 90.7 [75.2 to 150.2] | 87.6 [58.1 to 142.3] | 61.1 [50.5 to 76.2] | 54.1 [47.8 to 63.0] | 57.1 [50.6 to 69.0] | 128.6 [90.7 to 156.8] | 59.1 [47.3 to 73.5] | 125.1 [93.0 to 188.2]

2. Primary Outcome: Percent Change of E1, E2, and E1S Levels at 9, 10.5, and 12 Months From Baseline, by Treatment Group
Description: Changes in hormone levels (E1, E2, and E1S levels), as percentage change over time according to treatment assignment (at 9, 10.5 and 12 months from baseline).
Time Frame: 9, 10.5, and 12 months from baseline
Population: Longitudinal Analysis Population: There were 90/103 patients (21 continuous, 69 intermittent) who had baseline and one or more samples at 9, 10.5 and/or 12 months and could be included in analyses of hormone levels over time. 90 patients at baseline, 85 patients at month 9, 84 patients at month 10.5, and 81 patients at month 12.
Measure: Median (Inter-Quartile Range); unit: percentage change
Groups:
- Continuous Letrozole Treamtnet Group (9 Months): There were 90/103 patients (21 continuous, 69 intermittent) who had baseline and one or more samples at 9, 10.5 and/or 12 months and could be included in analyses of hormone levels over time. At 9, 10.5, and 12 months, 85 (21 continuous, 64 intermittent)/, 84 (20 continuous, 64 intermittent), and 81 (19 continuous, 62 intermittent), patients, respectively, could be included in analyses of hormone levels over time.
- Continuous Letrozole Treatment Arm (10.5 Months); Intermittent Letrozole Treatment Group (10.5 Months); Continuous Letrozole Treatment Arm (12 Months); Intermittent Letrozole Treatment Group (12 Months): There were 90/103 patients (21 continuous, 69 intermittent) who had baseline and one or more samples at 9, 10.5 and/or 12 months and could be included in analyses of hormone levels over time. At 9, 10.5, and 12 months, 85 (21 continuous, 64 intermittent), 84 (20 continuous, 64 intermittent), and 81 (19 continuous, 62 intermittent), patients, respectively, could be included in analyses of hormone levels over time.
Arm/Group | Continuous Letrozole Treamtnet Group (9 Months) | Intermittent Letrozole Treatment Group (9 Months) | Continuous Letrozole Treatment Arm (10.5 Months) | Intermittent Letrozole Treatment Group (10.5 Months) | Continuous Letrozole Treatment Arm (12 Months) | Intermittent Letrozole Treatment Group (12 Months)
Number analyzed (Participants) | 21 | 64 | 20 | 64 | 19 | 62
percentage change
  Percent change of E1 | -58.2 [-77.2 to -44.9] | -59.3 [-79.4 to -13.9] | -67.3 [-81.1 to -53.0] | 76.6 [-22.7 to 289.3] | -57.8 [-75.4 to -34.8] | 68.7 [-14.4 to 318.9]
  Percent change of E2 | -34.2 [-59.2 to -10.6] | -32.2 [-58.9 to -2.8] | -39.6 [-56.9 to -11.1] | 62.7 [-18.1 to 111.3] | -47.7 [-60.5 to 0.2] | 46.2 [-12.1 to 118.3]
  Percent change of ES1: number analyzed (Participants) | 21 | 63 | 20 | 63 | 19 | 62
  Percent change of ES1 | -29.8 [-60.9 to -15.3] | -42.3 [-62.2 to -7.9] | -38.7 [-63.4 to -22.6] | 32.9 [-20.3 to 96.7] | -36.7 [-68.5 to -21.5] | 31.6 [-2.4 to 103.1]

3. Secondary Outcome: Toxicity Grade Changes for Arthralgia, Hot Flushes, and Insomnia
Description: Toxicity grade changes from 6 to 12 months (hot flashes, insomnia and arthralgia; Common Terminology Criteria for Adverse Events (CTCAE) version 3 values 1- 4 grouped as no change, increase in grade [worsening] or decrease in grade [improvement])
Time Frame: 6 and 12 months
Population: In total, 76/85 patients (19 continuous; 57 intermittent) who had a 9 month sample also had a sample at 12 months and are included in analyses relating E2 change (9 to 12m) with QL, grip strength and adverse event (AE) changes.
Measure: Median (Inter-Quartile Range); unit: toxicity grade
Groups:
- Continuous Letrozole Treatment Group; Intermittent Letrozole Treatment Group: In total, 76/85 patients (19 continuous; 57 intermittent) who had a 9 month sample also had a sample at 12 months and are included in analyses relating E2 change (9 to 12m) with QL, grip strength and AE changes.
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Number analyzed (Participants) | 19 | 57
toxicity grade
  AE: Hot Flushes Grade Change from 6 to 12 Months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  AE: Insomnia Grade Change from 6 to 12 Months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  AE: Arthralgia Grade Change from 6 to 12 Months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Quality of Life (QoL) Score Changes
Description: All patients in SOLE-EST were assessed for symptom specific QoL. QoL changes from 6 to 12 months (sleep change, hot flushes, tiredness, difficulties of becoming aroused, loss of sexual interest, physical wellbeing and mood; LASA (linear analogue self-assessment) scores 0-100 (higher is better QoL) were calculated as 12 months minus 6 months, so that negative is worsening and positive is improvement.
Time Frame: 6 and 12 months: Change is calculated from 12 months minus 6 months, therefore positive values indicate an improved condition and negative values indicate a declined condition
Population: In total, 76/85 patients (19 continuous; 57 intermittent) who had a 6 month sample also had a sample at 12 months and are included in analyses relating E2 change (6 to 12m) with QL, grip strength and AE changes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Continuous Letrozole Treatment Group; Intermittent Letrozole Treatment Group: In total, 76/85 patients (19 continuous; 57 intermittent) who had a 6 month sample also had a sample at 12 months and are included in analyses relating E2 change with quality of life.
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Number analyzed (Participants) | 19 | 57
score on a scale
  LASA sleep disturbance score change from 12 to 6 months: number analyzed (Participants) | 16 | 54
  LASA sleep disturbance score change from 12 to 6 months | 0.0 [-6.5 to 14.5] | -9.5 [-27.0 to 2.0]
  LASA hot flush score change from 12 to 6 months: number analyzed (Participants) | 17 | 53
  LASA hot flush score change from 12 to 6 months | 2.0 [-3.0 to 12.0] | -2.0 [-13.0 to 6.0]
  LASA tiredness score change from 12 to 6 months: number analyzed (Participants) | 17 | 55
  LASA tiredness score change from 12 to 6 months | -1.0 [-19.0 to 7.0] | -9.0 [-23.0 to 3.0]
  LASA difficulty becoming aroused score change from 12 to 6 months: number analyzed (Participants) | 8 | 25
  LASA difficulty becoming aroused score change from 12 to 6 months | 0.5 [-7.5 to 20.5] | 0.0 [-16.0 to 3.0]
  LASA loss of sexual interest score change from 12 to 6 months: number analyzed (Participants) | 13 | 44
  LASA loss of sexual interest score change from 12 to 6 months | -3.0 [-18.0 to 8.0] | -1.5 [-8.5 to 4.5]
  LASA physical well-being score change from 12 to 6 months: number analyzed (Participants) | 16 | 55
  LASA physical well-being score change from 12 to 6 months | -1.0 [-13.5 to 5.5] | -5.0 [-19.0 to 12.0]
  LASA mood score change from 12 to 6 months: number analyzed (Participants) | 17 | 55
  LASA mood score change from 12 to 6 months | 0.0 [-3.0 to 7.0] | -1.0 [-24.0 to 10.0]

5. Secondary Outcome: Change in Grip-strength Score in the Dominant Hand
Description: Grip strength was measured using the Martin Vigorimeter (a modified sphygmomanometer which measures the force of compression in kilo pascal by means of a compressible rubber ball). To perform the hand grip test, the patients were asked to squeeze the ball of a modified sphygmomanometer three times with maximal force and the maximal value of three trials of each hand were used for evaluation. Higher value represents greater strength, thus changes are calculated as 12 months minus 9 months so that positive is improved condition and negative is declined condition.
Time Frame: Changes in grip strength score is calculated at 12 months minus 9 months
Population: Longitudinal analysis population N=90 (21 Continuous letrozole; 69 Intermittent letrozole); N samples per timepoint: N=90 at baseline, N=85 at month 9; N= 84 at month 10.5, N=81 at month 12. In total, 76/85 patients (19 continuous; 57 intermittent) who had a 9 month sample also had a sample at 12 months and are included in analyses relating E2 change (9 to 12m) with grip strength.
Measure: Median (Inter-Quartile Range); unit: kilopascals
Groups:
- Continuous Letrozole Treatment Group; Intermittent Letrozole Treatment Group: Longitudinal analysis population N=90 (21 Continuous letrozole; 69 Intermittent letrozole); N samples per timepoint: N=90 at baseline, N=85 at month 9; N= 84 at month 10.5, N=81 at month 12. In total, 76/85 patients (19 continuous; 57 intermittent) who had a 9 month sample also had a sample at 12 months and are included in analyses relating E2 change (9 to 12m) with QL, grip strength and AE changes.
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
Number analyzed (Participants) | 19 | 57
kilopascals | -1.0 [-6.0 to 2.0] | 0.0 [-6.0 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) information were collected at baseline and at 6 and 12 months in the SOLE main study.
Description: Adverse event (AE) information were collected at baseline and at 6 and 12 months in the SOLE main study, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v3.0). Primary AEs for the SOLE-EST substudy are arthralgia, hot flushes and insomnia (reported in the results module).
Arm/Group | Continuous Letrozole Treatment Group | Intermittent Letrozole Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/78
Other Adverse Events (participants affected / at risk) | 0/25 | 0/78

LIMITATIONS AND CAVEATS:
After 5 years of adjuvant endocrine therapy, resistant tumoral cells could be different from those present at initial diagnosis, and the apoptotic effect of estrogen on these cells might be insufficient. It is possible that the intermittent treatment was given too late.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-07-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT01281137/Prot_SAP_000.pdf